CLINICAL TRIAL: NCT06661486
Title: Evidence-based Lifestyle Interventions for the Delay of Cognitive Decline Among Older Singaporeans: Cohort Study and Randomized Controlled Trial
Brief Title: Evidence-based Lifestyle Interventions for the Delay of Cognitive Decline Among Older Singaporeans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Feng Lei, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NUS-IRB-2023-219; MOH-001290 (Other Grant/Funding Number: National Medical Research Council)
Record Dates: First submitted 2024-06-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-06

CONDITIONS: Non Demented
Keywords: Lifestyle Intervention; MMSE; CDR

STUDY DESIGN:
Intervention Model Description: the participants will be randomly assigned to one of the three arms, uniformed intervention, individualized intervention or the control group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): The control group will not receive any intervention and, is only required to attend 3 timepoints of cognitive assessment: baseline, 12 months and 24 months.
- Uniformed intervention group (Experimental): Uniformed intervention groups receive health education sessions in a group setting. Each session is one hour, and lifestyle health-related topics will be delivered to the participants for their knowledge.
  Interventions: Behavioral: Uniformed intervention group
- Individualised intervention group (Active Comparator): The individualised intervention group receives health education sessions as the uniformed intervention group and receives additional one-on-one health coaching, which besides the group sessions, the participants receive individual sessions every three months.
  Interventions: Behavioral: Individualised intervention group

INTERVENTIONS:
Behavioral: Uniformed intervention group — The investigators provide lifestyle intervention through a health education programme which is in a group setting. The sessions consisted of short talks on a health-related topic targeting lifestyle factors associated with dementia risk, followed by group activities that required interactions, cognitive engagement, and the acquisition of certain skills (for example, how to read food labels, how to measure blood pressure, how to recognize signs of depression, et al).
  Arms: Uniformed intervention group
Behavioral: Individualised intervention group — On top of the uniformed intervention group, the individualised intervention group receives also 1:1 sessions every 3 months within 2 years. Participants will review the knowledge taught in the group sessions individually and the investigator will address the participant's concerns and provide advice to the participant for a better lifestyle accordingly.
  Arms: Individualised intervention group

SUMMARY:
The investigators aim to investigate the relationship between lifestyle factors and cognitive decline among older Singaporeans and assess the feasibility and preliminary efficacy of a lifestyle intervention programme in delaying cognitive decline. Healthy lifestyle is a way of living that can lower down disease risk and promote health and wellbeing. Accumulating evidences support that lifestyle factors contribute to the development of dementia and hence modifying lifestyle could be a promising approach for dementia prevention. The intervention will focus on the promotion of a brain-healthy lifestyle, with special attention paid to common problems among local older adults. The investigators will assess cognitive and biological changes using the following outcome measures. Primary outcome: the processing speed domain Z score derived from raw scores of three tests including the symbol digit modality test, Colour trial test, and Stroop test (condition 2). Secondary outcome: i. epigenetic age (DNA methylation), ii. plasma-based markers of inflammation, iii. activities of daily living and instrumental activities of daily living, iv. Health-related quality of life measured by the EQ-5D-5L scale, v. wellbeing measured by the ICECAP-O (ICEpop CAPability measure for Older people), vi. other neurocognitive assessment tests. The investigators hypothesize that:

1. Lifestyle factors are associated with cognitive decline, epigenetic age, and systematic chronic inflammation.
2. Evidence-based lifestyle intervention focusing on common problems among local population can delay cognitive decline, slow epigenetic ageing, and produce favorable changes on chronic systemic inflammation.
3. Changes in biological markers will correlate with changes in cognitive function, and hence partially explains the observed clinical efficacy.
4. The interventions may also improve daily functioning, health-related quality of life, and wellbeing.
5. Interventions delivered in an individualized manner would produce more benefits than interventions delivered uniformly without considering individual's risk profile and personal and social context.

DETAILED DESCRIPTION:
The investigators have 3 arms in the trial, control group, uniformed intervention group, and individualised intervention group. The control group will not receive any intervention, while the intervention groups will receive group-based health education for 2 years. Within the 2 years, the health education will be conducted weekly in group-setting during the first month, and monthly on the months to follow. It will consist of short-talks on health-related topics that promote the lifestyle factors. Participants in individualized intervention group will undergo one-on-one health coaching session for every 3 months in addition to the group sessions. These will primarily serve to review what has been taught during the group interventions, and help the participants in addressing any questions and concerns they may have.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 60-75 years;
* (2) Singapore Modified Mini-Mental State Examination total score lower than locally validated education-specific cutoffs: < 25, 27 and 29 for those with nil, primary and secondary school and above education levels, respectively66.
* (3) Non-demented (Clinical Dementia Rating global score = 0).

Exclusion Criteria:

Conditions preventing effective engagement in the intervention

* (1) Terminal illness, aphasia
* (2) Marked hearing impairment
* (3) Participation in another interventional study

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Standard Neuropsychological Tests of Information Processing Speed | Cognitive assessment will be conducted at three timepoints within 2 years period, baseline, 12 months and 24 months
  The primary outcome of the trial is the processing speed, measured using the average of domain Z score derived from raw scores of three tests including the symbol digit modality test, colour trial test (Condition A) and Stroop test (Condition 2). The average of Z scores standardised to the baseline mean and standard deviation of trial participants, with higher scores representing better processing speed.

SECONDARY OUTCOMES:
Biological Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Secondary outcome measures include biological outcome: i. epigenetic age (DNA methylation)
Biological Outcome | All of the outcome meausures will be measured at three timepoints including baseline, 12 months and 24 months
  Secondary outcome measures include biological outcome: ii. plasma-based markers of inflammation
Quality of life Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Health-related Quality-of-life questionnaires: EuroQol-5 Dimension 5 Levels EQ-5D-5L. The result will not derive a summary score, "1" represents no problem and "5" represents extreme.
Quality of life Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Quality-of-life questionnaires: ICEpop CAPability measure for Older adults ICECAP-O. The result will not derive a summary score, "1" represents no ability, "4" represents no problem.
Social Support Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Duke Social Support Index DSSI-11. The sum of 11 items, a higher score represents better social support. Minimum 11, maximum 33.
Capability-related Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Capability-related questionnaires: Basic Activities of Daily Living ADL The sum of 10 items. A higher score represents better capability: minimum 0, maximum 20.
Capability-related Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Capability-related questionnaires: Instrumental Activities of Daily Living IADL.The sum of 8 items, a higher score represents better capability: minimum 0, maximum 8.
Sleep Quality Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Pittsburgh Sleep Quality Index PSQI. A sum of 7 components, with global scores ranging from 0-21, a higher score represents worse sleep quality.
Mental Health Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Mental health outcome: Geriatric Depression Scale GDS. A sum score of 15 items, a lower score represents lesser depression: Minimum 0, maximum 15.
Mental Health Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Mental health outcome: Geriatric Anxiety Inventory GAI. A sum score of 20 items, a lower score represents lesser anxiety: Minimum 0, maximum 20.
Mental Health Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Mental health outcome: Perceived Stress Scale PSS. A sum score of 10 items, a lower score represents lower stress: Minimum 0, maximum 40.
Cognitive Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Mini-Mental State Examination (MMSE), total score of 30 items, a higher score better cognitive: Minimum 0, maximum 30.
Cognitive Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Clinical Dementia Rating (CDR), a higher score higher impairment in cognitive function, high risk in dementia, global score ranged from 0 to 3.
Neurocognitive Tests Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Neuropsychological tests: Rey Auditory Verbal Learning Test (RAVLT). Different summary scores are derived from raw RAVLT scores: Minumum 0, maximum 15. A higher score better verbal memory.
Neurocognitive Tests Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Neuropsychological tests: Digit Span Task. Higher scores represent better cognitive performance.
Neurocognitive Tests Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Neuropsychological test: Block Design (BD). Higher scores represent better cognitive performance: Minimum 0, Maximum 68.
Neurocognitive Tests Outcome | All of the outcome measures will be measured at three timepoints including baseline, 12 months and 24 months
  Neuropsychological test: Boston Naming Test (BNT) . Higher scores represent better cognitive performance: Minimum 0, maximum 30.

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - National University Singapore, Tahir Foundation Building, Singapore, Singapore
  - National University Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu LY, Lu Y, Shen L, Li CB, Yu JT, Yuan CR, Ye KX, Chao YX, Shen QF, Mahendran R, Kua EH, Yu DH, Feng L. Prevalence, risk and protective factors for mild cognitive impairment in a population-based study of Singaporean elderly. J Psychiatr Res. 2022 Jan;145:111-117. doi: 10.1016/j.jpsychires.2021.11.041. Epub 2021 Nov 25. PMID 34894520
- [Background] Ye KX, Sun L, Wang L, Khoo ALY, Lim KX, Lu G, Yu L, Li C, Maier AB, Feng L. The role of lifestyle factors in cognitive health and dementia in oldest-old: A systematic review. Neurosci Biobehav Rev. 2023 Sep;152:105286. doi: 10.1016/j.neubiorev.2023.105286. Epub 2023 Jun 13. PMID 37321363
- [Background] Wu DX, Feng L, Yao SQ, Tian XF, Mahendran R, Kua EH. The early dementia prevention programme in Singapore. Lancet Psychiatry. 2014 Jun;1(1):9-11. doi: 10.1016/S2215-0366(14)70233-0. Epub 2014 Jun 4. No abstract available. PMID 26360390